CLINICAL TRIAL: NCT02904707
Title: Interest of Skin Graft Pellets in the Management of Ulcers Algic
Acronym: ULCERALGIQUE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ULCERALGIQUE
Record Dates: First submitted 2016-09-01; First posted 2016-09-19 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2016-09

CONDITIONS: Ulcer, Leg; Ulcer Algic
Keywords: Skin Graft
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionary EQ-5D: The EQ-5D questionary will be distributed at the beginning of hospitalization and completed by each patient, and will evaluate the impact of painful ulcers in their daily lives.
  Finally, a pain assessment questionnaire by Numeric Evaluation Scale before and after the skin graft pellet, will be filled by a caregiver during an interview with each patient.
  Interventions: Other: Questionary EQ-5D

INTERVENTIONS:
Other: Questionary EQ-5D — In addition to the pain questionary that is filled filled as usual, the EQ-5D questionary will be distributed at the beginning of hospitalization and completed by each patient, and will evaluate the impact of painful ulcers in their daily lives.

SUMMARY:
Leg ulcers (UDJ) is defined as a chronic skin wound, lasting for more than 4 to 6 weeks, between the knee and foot, and with no tendency to spontaneous healing.

In 2002, the prevalence of leg ulcers is estimated between 0.5% and 1% of the general population and 3% in subjects over 65 years.

The sex ratio is generally 3 females to 1 male. It is in most cases a complication of vascular disease, usually venous (70 to 90%), then blood (5-15%), mixed (5-10%) and microcirculatory.

In three quarter of cases, the UDJ is a chronic painful wound to the social repercussions (sleep disorders, eating, work stoppages) and major economic (individual and collective costs of absorptions).

The treatment of a chronic wound uses validated techniques for several years as the skin graft in tablets, associated with the etiological treatment.

The latest recommendations HAS implemented to date from 2006 and concerns the management of leg ulcers predominantly venous.

Few articles in the literature address the possibility of an analgesic effect of the transplant pellets in the treatment of chronic ulcers algic.

In 2008, a Swedish article, evaluated pain before and after skin grafting in carriers of leg ulcer patients and feet and showed that there was a reduction in pain post transplant.

We propose to evaluate the analgesic effect of the skin graft in pellet on a patient population having one or more Algic ulcers.

DETAILED DESCRIPTION:
Development of the study:

An information note and the non-opposition of the patient will be collected on the first day of hospitalization. The written and signed consent will be recorded in the patient record.

Clinical data will be collected during hospitalization of the patient, respecting his anonymity only initials and year of birth will be made in terms of data that distinguish patients.

The EQ-5D questionary will be distributed at the beginning of hospitalization and completed by each patient, and will evaluate the impact of painful ulcers in their daily lives.

Finally, a pain assessment questionary by NE (Numeric Evaluation) before and after the skin graft pellet, will be filled by a caregiver during an interview with each patient.

Methodology :

Design: open, prospective, single centric (Vascular Medicine Department), Interventional.

The data to be collected are:

The age, sex, weight, height Length of hospitalization, The type of ulcer, the size of the ulcer disease duration of current or ulcers, duration of ulcer disease The graft antecedent, number of grafts placed in the registry, the date of completion of the graft, The evaluation of pain before and after the completion of the graft on EN, The impact of pain on patient's quality of sleep, the type of pain experienced by patients in terms of their ulcers

The type and number of analgesics taken by patients:

* Antiepileptic therapy (pregabapentine, gabapentin)
* Analgesic treatment to alleviate I (paracetamol), to overcome II (codeine paracetamol, Lamaline, tramadol, nefopam, Ixprim), and compensate III (morphine, opiates).

ELIGIBILITY:
Inclusion Criteria:

* Inpatient consecutively
* over 18 years old, man, woman,
* having one or more ulcers of venous, arterial or microcirculatory
* for more than four to six weeks
* answering yes to the question: is it painful ulcer?
* consultant in vascular medicine department of St. Joseph hospital in February the month of April 2015

Exclusion Criteria:

* Patients minors
* Patients with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with one or more ulcers of venous, arterial or microcirculatory origin for more than four to six weeks
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of change of pain by Numeric Evaluation Scale | Day -1, Day 1 and Day 7
  A pain assessment questionnaire by Numeric Evaluation Scale NE (pain rating scale measuring pain intensity from 0 to 10) before and after the skin graft pellet, will be filled by a caregiver during an interview with each patient

SECONDARY OUTCOMES:
Assessment of change of the impact of painful ulcers usin EQ-5D Questionary | Day -1, Day 1 and Day 7
  The EQ-5D questionnaire will be distributed at the beginning of hospitalization and completed by each patient, and will evaluate the impact of painful ulcers in their daily lives.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAZARETH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided